CLINICAL TRIAL: NCT01807221
Title: A Randomized, Double-blind, Double-dummy, Multi-center Study to Assess Safety and Efficacy of Different Oral Doses of BAY94-8862 in Subjects With Emergency Presentation at the Hospital Because of Worsening Chronic Heart Failure With Left Ventricular Systolic Dysfunction and Either Type 2 Diabetes Mellitus With or Without Chronic Kidney Disease or Chronic Kidney Disease Alone Versus Eplerenone
Brief Title: Phase IIb Safety and Efficacy Study of Different Oral Doses of BAY94-8862 in Subjects With Worsening Chronic Heart Failure and Left Ventricular Systolic Dysfunction and Either Type 2 Diabetes Mellitus With or Without Chronic Kidney Disease or Chronic Kidney Disease Alone
Acronym: ARTS-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14564; 2012-002627-15 (EudraCT Number)
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Heart Decompensation
MeSH Terms: conditions — Heart Failure | interventions — finerenone; Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Finerenone(BAY94-8862)[2.5mg] + Placebo (Experimental): Oral - 2.5mg once daily (OD) for 30 days. Potential up-titration to 5mg OD after 30 days or 60 days. Treatment duration 90 days. Placebo OD for 90 days.
  Interventions: Drug: Finerenone (BAY94-8862); Drug: Placebo
- Finerenone (BAY94-8862)[5mg] + Placebo (Experimental): Oral - 5mg OD for 30 days. Potential up-titration to 10 mg OD after 30 days or 60 days. Treatment duration 90 days. Placebo OD for 90 days.
  Interventions: Drug: Finerenone (BAY94-8862); Drug: Placebo
- Finerenone (BAY94-8862)[7.5mg] + Placebo (Experimental): Oral - 7.5mg OD for 30 days. Potential up-titration to 15 mg OD after 30 days or 60 days. Treatment duration 90 days. Placebo OD for 90 days.
  Interventions: Drug: Finerenone (BAY94-8862); Drug: Placebo
- Finerenone (BAY94-8862)[10mg] + Placebo (Experimental): Oral - 10mg OD for 30 days. Potential up-titration to 20 mg OD after 30 days or 60 days. Treatment duration 90 days. Placebo OD for 90 days.
  Interventions: Drug: Finerenone (BAY94-8862); Drug: Placebo
- Finerenone (BAY94-8862)[15mg] + Placebo (Experimental): Oral - 15mg OD for 30 days. Potential up-titration to 20 mg OD after 30 days or 60 days. Treatment duration 90 days. Placebo OD for 90 days.
  Interventions: Drug: Finerenone (BAY94-8862); Drug: Placebo
- Eplerenone [25 mg] + Placebo (Active Comparator): Oral - 25mg every other day (EOD). Potential up-titration to 25mg OD after 30 days and 50mg OD after 60 days.Placebo OD for 90 days.
  Interventions: Drug: Placebo; Drug: Inspra (eplerenone)

INTERVENTIONS:
Drug: Finerenone (BAY94-8862)
  Arms: Finerenone (BAY94-8862)[10mg] + Placebo; Finerenone (BAY94-8862)[15mg] + Placebo; Finerenone (BAY94-8862)[5mg] + Placebo; Finerenone (BAY94-8862)[7.5mg] + Placebo; Finerenone(BAY94-8862)[2.5mg] + Placebo
Drug: Placebo
Drug: Inspra (eplerenone)
  Arms: Eplerenone [25 mg] + Placebo

SUMMARY:
To assess a new drug, BAY94-8862, given orally at different doses, to evaluate whether it was safe and can help the well-being of patients with worsening chronic heart failure and either type II diabetes with or without chronic kidney disease or kidney disease alone. These treatment doses were compared to eplerenone, another marketed drug approved to treat heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older. The lower age limit may be higher if legally required in the participating country
* Women of childbearing potential can only be included in the study if a pregnancy test is negative and if they agree to use adequate contraception when sexually active
* Subjects with worsening chronic heart failure requiring emergency presentation to hospital and treatment with intravenous diuretics at hospital
* Subjects with clinical diagnosis of chronic heart failure (CHF) either ischemic or non ischemic, New York Heart Association (NYHA) functional class II-IV
* Subjects with type 2 diabetes mellitus and / or
* Subjects with 30 mL/min/1.73m^2 </= eGFR </= 60 mL/min/1.73m^2 (MDRD, Modification of Diet in Renal Disease Study Group) at screening
* Left ventricular ejection fraction (LVEF) </= 40%
* Blood potassium </= 5.0 mmol/L at screening
* Systolic blood pressure >/= 90 mmHg without signs and symptoms of hypotension at the screening visit

Exclusion Criteria:

* Acute de-novo heart failure or acute inflammatory heart disease, e.g. acute myocarditis
* Acute coronary syndrome (ACS) in last 30 days prior to screening
* Cardiogenic shock
* Valvular heart disease requiring surgical intervention during the course of the study
* Stroke or transient ischemic cerebral attack in the last 3 months prior to the screening visit
* Concomitant treatment with any mineralocorticoid receptor antagonist (MRA), renin inhibitor, or potassium-sparing diuretic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1066 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2014-11-11 (Actual); Study Completion 2014-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (146):
- United States (9):
  - Birmingham, Alabama
  - La Jolla, California
  - Los Angeles, California
  - Jacksonville, Florida
  - Macon, Georgia
  - Baltimore, Maryland
  - Detroit, Michigan
  - Newark, New Jersey
  - Fairfield, Ohio
- Australia (4):
  - Darlinghurst, New South Wales
  - Adelaide, South Australia
  - Concord
  - Prahran
- Austria (6):
  - Krems, Lower Austria
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz, Upper Austria
  - Salzburg
  - Vienna
- Bulgaria (5):
  - Burgas
  - Pazardzhik
  - Rousse
  - Sofia
  - Varna
- Canada (7):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
  - Sherbrooke, Quebec
  - Québec
- Czechia (4):
  - Jindřichův Hradec
  - Ostrava
  - Prague
  - Slaný
- Denmark (10):
  - Copenhagen Ø
  - Esbjerg
  - Glostrup Municipality
  - Hellerup
  - Herlev
  - Hvidovre
  - København NV
  - Køge
  - Svendborg
  - Viborg
- Finland (4):
  - Espoo
  - Helsinki
  - Rovaniemi
  - Turku
- France (6):
  - Bron
  - Nice
  - Paris
  - Rouen
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (11):
  - Würzburg, Bavaria
  - Frankfurt am Main, Hesse
  - Limburg an der Lahn, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Stade, Lower Saxony
  - Bad Oeynhausen, North Rhine-Westphalia
  - Mönchengladbach, North Rhine-Westphalia
  - Homburg, Saarland
  - Erfurt, Thuringia
  - Berlin
- Greece (4):
  - Athens
  - Chaïdári
  - Larissa
  - Nea Ionia / Athens
- Hungary (3):
  - Budapest
  - Nagykanizsa
  - Székesfehérvár
- Israel (12):
  - Afula
  - Ashkelon
  - Hadera
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Rehovot
  - Safed
  - Tel Aviv
  - Ẕerifin
- Italy (8):
  - Foggia, Apulia
  - Rome, Lazio
  - Bergamo, Lombardy
  - Milan, Lombardy
  - Monza Brianza, Lombardy
  - Arezzo, Tuscany
  - Pisa, Tuscany
  - Perugia, Umbria
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Vilnius
- Netherlands (8):
  - Amsterdam
  - Delft
  - Groningen
  - Hoogeveen
  - Nijmegen
  - Rotterdam
  - Veldhoven
  - Zutphen
- Stavanger, Norway
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Gdansk
  - Katowice
  - Kielce
  - Krakow
  - Szczecin
  - Warsaw
  - Wroclaw
- Portugal (4):
  - Almada
  - Faro
  - Lisbon
  - Porto
- South Africa (9):
  - Petoria, Gauteng
  - Isipingo Rail, KwaZulu-Natal
  - Merebank, KwaZulu-Natal
  - Tongaat, KwaZulu-Natal
  - Cape Town, Western Cape
  - Kuils River, Western Cape
  - Pinelands, Western Cape
  - Somerset West, Western Cape
  - Worcester, Western Cape
- South Korea (2):
  - Wŏnju, Gang''weondo
  - Seoul
- Spain (6):
  - Olot, Girona
  - Majadahonda, Madrid
  - El Palmar, Murcia
  - Barcelona
  - Madrid
  - Valencia
- Sweden (5):
  - Falun
  - Gothenburg
  - Örebro
  - Stockholm
  - Umeå
- Taiwan (3):
  - New Taipei City
  - Taipei
  - Taizung
- Turkey (Türkiye) (3):
  - Ankara
  - Antalya
  - Izmir

REFERENCES:
- [Result] Filippatos G, Anker SD, Bohm M, Gheorghiade M, Kober L, Krum H, Maggioni AP, Ponikowski P, Voors AA, Zannad F, Kim SY, Nowack C, Palombo G, Kolkhof P, Kimmeskamp-Kirschbaum N, Pieper A, Pitt B. A randomized controlled study of finerenone vs. eplerenone in patients with worsening chronic heart failure and diabetes mellitus and/or chronic kidney disease. Eur Heart J. 2016 Jul 14;37(27):2105-14. doi: 10.1093/eurheartj/ehw132. Epub 2016 Apr 29. PMID 27130705
- [Result] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592
- [Result] Pitt B, Anker SD, Bohm M, Gheorghiade M, Kober L, Krum H, Maggioni AP, Ponikowski P, Voors AA, Zannad F, Nowack C, Kim SY, Pieper A, Kimmeskamp-Kirschbaum N, Filippatos G. Rationale and design of MinerAlocorticoid Receptor antagonist Tolerability Study-Heart Failure (ARTS-HF): a randomized study of finerenone vs. eplerenone in patients who have worsening chronic heart failure with diabetes and/or chronic kidney disease. Eur J Heart Fail. 2015 Feb;17(2):224-32. doi: 10.1002/ejhf.218. PMID 25678098
- [Derived] Ostrominski JW, Filippatos G, Claggett BL, Miao ZM, Desai AS, Jhund PS, Henderson A, Rohwedder K, Brinker MD, Scalise A, Schloemer P, Lam CSP, Senni M, Shah SJ, Voors AA, Zannad F, Rossing P, Ruilope LM, Anker SD, Pitt B, Agarwal R, McMurray JJV, Solomon SD, Vaduganathan M. Effect of Finerenone on Morbidity and Mortality in CKD. J Am Soc Nephrol. 2025 Sep 12. doi: 10.1681/ASN.0000000823. Online ahead of print. No abstract available. PMID 40938666
- See also: Click here to find results for studies related to Bayer Healthcare products. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 168 study centers in 25 countries worldwide, from 17 June 2013 (first participant first visit) to 09 December 2014 (last participant last visit).
Pre-assignment Details: Out of 1286 screened participants, 1066 participants were randomized, 1055 participants received study treatment and were valid for safety analysis set.
Groups:
- Eplerenone (INSPRA®): Eplerenone 25 milligram (mg) capsule every other day (EOD), on Day 1, Day 3, Day 5, etc, along with placebo capsule (matched to Eplerenone capsule) on Day 2, Day 4, Day 6, etc., and placebo tablet (matched to Finerenone tablet) once daily (OD).The dose could be increased to 25 mg OD at Day 30 and to 50 mg OD at Day 60 (or 25 mg OD if no up-titration occurred on Day 30) if both up-titration steps were performed. Treatment duration was for 90 days.
- Finerenone (BAY94-8862) 2.5-5 mg OD: Finerenone 2.5 mg immediate-release (IR) tablets OD and placebo capsule (matched to Eplerenone capsule) OD, with possible up-titration to 5 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
- Finerenone (BAY94-8862) 5-10 mg OD: Finerenone 5 mg IR tablets OD and placebo capsule (matched to Eplerenone capsule) OD, with possible up-titration to 10 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
- Finerenone (BAY94-8862) 7.5-15 mg OD: Finerenone 7.5 mg IR tablet OD and placebo capsule (matched to Eplerenone capsule) OD, with possible up-titration to 15 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
- Finerenone (BAY94-8862) 10-20 mg OD: Finerenone 10 mg IR tablet OD and placebo capsule (matched to Eplerenone capsule) OD, with possible up-titration to 20 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
- Finerenone (BAY94-8862) 15-20 mg OD: Finerenone 15 mg IR tablet OD and placebo capsule (matched to Eplerenone capsule) OD, with possible up-titration to 20 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
Period: Overall Study
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Started | 224 | 173 | 165 | 169 | 170 | 165
Participants Received Study Treatment and Valid for Safety Analysis Set | 221 | 172 | 163 | 167 | 169 | 163
Completed | 144 | 121 | 122 | 123 | 134 | 124
Not Completed | 80 | 52 | 43 | 46 | 36 | 41
Not completed — Progressive disease | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 7 | 9 | 4 | 2 | 1 | 6
Not completed — Physician Decision | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 33 | 22 | 26 | 25 | 18 | 21
Not completed — Protocol Violation | 0 | 2 | 1 | 2 | 0 | 1
Not completed — Non-compliance | 1 | 2 | 0 | 1 | 0 | 0
Not completed — Logistical difficulties | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 33 | 15 | 8 | 14 | 16 | 13
Not completed — Sponsor decision | 2 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): all randomized participants who took at least one dose of study drug and with data after beginning of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD | Total
Number analyzed (Participants) | 221 | 172 | 163 | 167 | 169 | 163 | 1055
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.38 (9.92) | 72.53 (9.74) | 71.81 (10.55) | 69.27 (9.83) | 71.27 (10.27) | 69.2 (10.15) | 71.15 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 37 | 37 | 43 | 41 | 31 | 240
  Male | 170 | 135 | 126 | 124 | 128 | 132 | 815
Baseline BNP [Geometric Mean (Standard Deviation); unit: pg/ml] — B-type natriuretic peptide (BNP) levels in the blood are used for screening, diagnosis of acute chronic heart failure (CHF) and may be useful to establish prognosis in heart failure. Population: Participants with valid data for this baseline characteristic
  pg/ml
    number analyzed (Participants) | 203 | 156 | 151 | 156 | 158 | 155 | 979
    (all) | 594.290 (2.601) | 677.906 (2.637) | 574.245 (2.543) | 570.776 (2.741) | 606.080 (2.598) | 552.032 (2.698) | 594.732 (2.634)
Baseline NT-proBNP [Geometric Mean (Standard Deviation); unit: pg/ml] — N-terminal pro-B type natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute chronic heart failure (CHF) and may be useful to establish prognosis in heart failure. Population: Participants with valid data for this baseline characteristic
  pg/ml
    number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158 | 1002
    (all) | 4730.170 (2.938) | 4793.430 (3.084) | 4184.631 (3.093) | 3776.859 (3.395) | 4163.898 (2.734) | 3791.677 (3.013) | 4246.883 (3.040)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Relative Decrease in NT-proBNP of More Than 30% From Baseline to Day 90
Description: N-terminal pro-B type natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute and chronic heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Baseline and Day 90
Population: Full analysis set (FAS): all participants who the study drug, had baseline and at least one post-baseline NT-proBNP value or who died or experienced permanent (≥5 consecutive days) withdrawal of study drug after cardiovascular (CV) hospitalization or after emergency presentation for Worsening Chronic Heart Failure (WCHF)
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Percentage of participants | 37.2 (31.6) [31.6 to 43.1] | 30.9 (24.9) [24.9 to 37.4] | 32.5 (26.3) [26.3 to 39.2] | 37.3 (30.9) [30.9 to 44.1] | 38.8 (32.3) [32.3 to 45.5] | 34.2 (27.9) [27.9 to 40.9]
Statistical Analysis 1: Comparison: Eplerenone (INSPRA®) vs Finerenone (BAY94-8862) 2.5-5 mg OD; Estimates and two-sided 90% confidence intervals are provided for each treatment group and for the treatment differences πBi - πC. Clopper-Pearson confidence intervals were calculated for each treatment group, while for treatment differences the exact unconditional confidence limits were calculated; Test type: Other; p = 0.8771, Chi-squared; Mean Difference (Final Values) = -6.3, 90% CI 2-sided [-14.9 to 2.3]
Statistical Analysis 2: Comparison: Eplerenone (INSPRA®) vs Finerenone (BAY94-8862) 5-10 mg OD; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.7945, Chi-squared; Mean Difference (Final Values) = -4.7, 90% CI 2-sided [-13.4 to 4]
Statistical Analysis 3: Comparison: Eplerenone (INSPRA®) vs Finerenone (BAY94-8862) 7.5-15 mg OD; Estimates and two-sided 90% confidence intervals are provided for each treatment group and for the treatment differences πBi - πC. Clopper-Pearsonconfidence intervals were calculated for each treatment group, while for treatment differences the exact unconditional confidence limits were calculated; Test type: Other; p = 0.5, Chi-squared; Mean Difference (Final Values) = 0.1, 90% CI 2-sided [-8.5 to 8.8]
Statistical Analysis 4: Comparison: Eplerenone (INSPRA®) vs Finerenone (BAY94-8862) 10-20 mg OD; [analysis description as in outcome 1, analysis 3]; Test type: Other; p = 0.4225, Chi-squared; Mean Difference (Final Values) = 1.6, 90% CI 2-sided [-7.1 to 10.2]
Statistical Analysis 5: Comparison: Eplerenone (INSPRA®) vs Finerenone (BAY94-8862) 15-20 mg OD; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.6865, Chi-squared; Mean Difference (Final Values) = -3, 90% CI 2-sided [-11.7 to 5.7]

2. Secondary Outcome: Number of Participants With Death Due to Any Cause
Description: Death due to any cause include cardiovascular (CV) death and Non-CV death. Non-CV death was classified by 2 subcategories: non-malignant causes and malignant causes.
Time Frame: Day 30, Day 60, Day 90 and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Participants
  Day 30 | 6 | 5 | 1 | 1 | 0 | 2
  Day 60 | 7 | 7 | 3 | 2 | 0 | 4
  Day 90 | 9 | 10 | 4 | 4 | 1 | 5
  Follow-up | 15 | 16 | 7 | 11 | 2 | 8

3. Secondary Outcome: Number of Participants With Cardiovascular Hospitalization
Description: Hospitalizations were defined as any unplanned admission to hospital, i.e. completion of hospital admission procedures and one overnight [i.e. date change] stay or until the death of subject occurred. Hospitalizations and deaths were classified by 2 primary categories: CV and non-CV. The pre-specified subcategories for CV hospitalizations were as follows: 1. Worsening heart failure, 2.Acute myocardial infarction, 3. Arrhythmia, 4.Transient ischemic attack and stroke, 5. Other CV hospitalizations.
Time Frame: Day 30, Day 60, Day 90 and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Participants
  Day 30 | 28 | 23 | 14 | 8 | 7 | 15
  Day 60 | 43 | 33 | 23 | 21 | 15 | 23
  Day 90 | 45 | 35 | 26 | 29 | 22 | 28
  Follow-up | 56 | 43 | 38 | 36 | 27 | 34

4. Secondary Outcome: Number of Participants With Emergency Presentations for Worsening Chronic Heart Failure (WCHF)
Description: Emergency presentations for WCHF were defined as newly developing signs and symptoms of WCHF after start of treatment with study drug, requiring an additional emergency presentation to hospital and IV treatment with diuretics and/or positive inotropic agents.
Time Frame: Day 30, Day 60, Day 90 and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Participants
  Day 30 | 21 | 19 | 12 | 9 | 7 | 15
  Day 60 | 35 | 30 | 20 | 17 | 14 | 22
  Day 90 | 37 | 32 | 22 | 24 | 18 | 28
  Follow-up | 47 | 40 | 30 | 30 | 26 | 34

5. Secondary Outcome: Ratio of BNP at Specified Visits to BNP at Baseline
Description: B-type natriuretic peptide (BNP) levels in the blood are used for screening, diagnosis of acute chronic heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: Day 30, Day 60, Day 90, Premature discontinuation (only for participants who have discontinued the study prematurely, to be performed as soon as possible after withdrawal of study drug) and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in FAS with valid data at specified visits
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 203 | 156 | 151 | 156 | 158 | 155
Ratio
  Day 30: number analyzed (Participants) | 176 | 136 | 136 | 141 | 139 | 133
  Day 30 | 0.925 (2.02) | 0.944 (1.952) | 0.878 (1.713) | 0.832 (1.959) | 0.852 (1.901) | 0.879 (1.968)
  Day 60: number analyzed (Participants) | 148 | 130 | 128 | 125 | 133 | 128
  Day 60 | 0.783 (2.194) | 0.864 (2.139) | 0.854 (1.854) | 0.79 (2.179) | 0.711 (2.116) | 0.824 (2.142)
  Day 90: number analyzed (Participants) | 141 | 119 | 122 | 119 | 127 | 120
  Day 90 | 0.723 (2.202) | 0.813 (2.412) | 0.839 (1.93) | 0.719 (2.204) | 0.706 (2.34) | 0.771 (2.197)
  Premature discontinuation: number analyzed (Participants) | 33 | 23 | 22 | 19 | 21 | 22
  Premature discontinuation | 0.896 (0.896) | 1.104 (2.15) | 1.006 (2.422) | 0.884 (1.973) | 0.848 (2.218) | 1.044 (2.174)
  Follow-up: number analyzed (Participants) | 165 | 128 | 136 | 126 | 143 | 136
  Follow-up | 0.795 (2.232) | 0.815 (2.388) | 0.886 (2.199) | 0.726 (2.397) | 0.729 (2.487) | 0.852 (2.169)

6. Secondary Outcome: Ratio of NT-proBNP at Specified Visits to NT-proBNP at Baseline
Description: N-terminal pro-B type natriuretic peptide (NT-proBNP) levels in the blood are used for screening, diagnosis of acute chronic heart failure (CHF) and may be useful to establish prognosis in heart failure.
Time Frame: as for outcome 5
Population: Participants in FAS with valid data at specified visits
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Ratio
  Day 30: number analyzed (Participants) | 177 | 137 | 139 | 145 | 141 | 136
  Day 30 | 0.883 (2.458) | 0.98 (2.158) | 0.874 (2.14) | 0.888 (2.123) | 0.822 (2.217) | 0.921 (2.136)
  Day 60: number analyzed (Participants) | 153 | 131 | 127 | 125 | 137 | 130
  Day 60 | 0.749 (2.73) | 0.822 (2.423) | 0.814 (2.178) | 0.81 (2.268) | 0.748 (2.496) | 0.829 (2.288)
  Day 90: number analyzed (Participants) | 142 | 119 | 120 | 118 | 129 | 121
  Day 90 | 0.688 (2.59) | 0.789 (2.661) | 0.765 (2.214) | 0.783 (2.454) | 0.728 (2.795) | 0.771 (2.471)
  Premature discontinuation: number analyzed (Participants) | 36 | 23 | 24 | 21 | 22 | 25
  Premature discontinuation | 0.948 (2.684) | 1.369 (2.087) | 1.267 (2.261) | 0.927 (1.864) | 1.133 (2.981) | 0.965 (2.352)
  Follow-up: number analyzed (Participants) | 165 | 130 | 139 | 131 | 144 | 137
  Follow-up | 0.747 (2.616) | 0.747 (2.741) | 0.887 (2.604) | 0.809 (2.647) | 0.746 (2.472) | 0.849 (2.348)

7. Secondary Outcome: Change From Baseline in KCCQ Questionnaire Scores at Specified Visits
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) was the leading health related quality of life measure for subjects with CHF. KCCQ was a 23 item questionnaire that independently measures the impact of subjects HF, or its treatment, on 7 distinct domains: self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ clinical summary score is a composite assessment of physical limitations and total symptom scores. Results from the total symptom summary score are presented. Scores are transformed to a range of 0-100, in which higher scores reflect better health status. In the below table, categorical data represents change from baseline data at respective time points.
Time Frame: Baseline, Day 30 and Day 90
Population: Participants in FAS with valid data at specified visits
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 203 | 161 | 156 | 158 | 160 | 157
Scores on a scale
  Baseline | 43.7 (23) | 42.8 (22.6) | 45.4 (24) | 42.1 (23.2) | 42.3 (23.7) | 43.2 (22.5)
  Day 30: number analyzed (Participants) | 177 | 141 | 137 | 145 | 141 | 141
  Day 30 | 20.5 (26.2) | 18.2 (22.7) | 19.3 (26.5) | 23 (24.4) | 24.9 (22.9) | 20.6 (27)
  Day 90: number analyzed (Participants) | 141 | 118 | 121 | 118 | 129 | 119
  Day 90 | 24.3 (27.6) | 21.3 (27.2) | 24.5 (27) | 29.3 (28.6) | 28.3 (23.8) | 22.2 (30.6)

8. Secondary Outcome: Change From Baseline in EQ-5D-3L Questionnaire Scores at Specified Visits
Description: EuroQol Group 5-Dimension, 3-Level (EQ-5D-3L): participant rated questionnaire to assess health-related quality of life. It consists of EQ-5D descriptive system and EQ-5D Visual Analog Scale (VAS). EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems (1), some problems (2), and extreme problems (3). For this population, the possible EQ-5D-3L index scores ranges from -0.11 (that is, 3 for all 5 dimensions) to 1.0 (that is, 1 for all 5 dimensions), where higher scores indicate a better health state.
Time Frame: Baseline, Day 30, Day 90, Premature discontinuation (only for participants who have discontinued the study prematurely, to be performed as soon as possible after withdrawal of study drug) and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in FAS with valid data at specified visits
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 207 | 162 | 157 | 158 | 160 | 158
Scores on scale
  Baseline: number analyzed (Participants) | 201 | 160 | 156 | 157 | 158 | 158
  Baseline | 0.58 (0.25) | 0.59 (0.25) | 0.62 (0.23) | 0.58 (0.23) | 0.56 (0.25) | 0.59 (0.24)
  Day 30: number analyzed (Participants) | 173 | 141 | 137 | 143 | 139 | 135
  Day 30 | 0.06 (0.23) | 0.02 (0.24) | 0.02 (0.23) | 0.07 (0.22) | 0.06 (0.23) | 0.02 (0.25)
  Day 90: number analyzed (Participants) | 139 | 117 | 122 | 117 | 126 | 120
  Day 90 | 0.08 (0.24) | 0.03 (0.27) | 0.04 (0.25) | 0.08 (0.2) | 0.1 (0.24) | 0.06 (0.28)
  Premature discontinuation: number analyzed (Participants) | 33 | 20 | 19 | 21 | 17 | 23
  Premature discontinuation | -0.12 (0.25) | -0.06 (0.29) | -0.09 (0.24) | -0.1 (0.24) | -0.05 (0.25) | 0 (0.29)
  Follow-up: number analyzed (Participants) | 161 | 129 | 136 | 133 | 144 | 139
  Follow-up | 0.06 (0.26) | 0.01 (0.25) | 0.01 (0.27) | 0.08 (0.23) | 0.07 (0.23) | 0.04 (0.28)

9. Other Pre Specified Outcome: Change From Baseline in Serum Potassium at Specified Visits
Time Frame: Baseline, Day 30, Day 60, Day 90 and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in SAF with valid data at specified visits
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 221 | 172 | 162 | 167 | 168 | 163
millimoles per liter (mmol/L)
  Baseline | 4.159 (0.495) | 4.081 (0.501) | 4.211 (0.541) | 4.174 (0.443) | 4.131 (0.506) | 4.117 (0.506)
  Day 30: number analyzed (Participants) | 178 | 136 | 137 | 142 | 143 | 137
  Day 30 | 0.057 (0.608) | 0.135 (0.573) | 0.075 (0.523) | 0.085 (0.475) | 0.21 (0.592) | 0.193 (0.556)
  Day 60: number analyzed (Participants) | 151 | 130 | 125 | 129 | 134 | 129
  Day 60 | 0.179 (0.589) | 0.091 (0.568) | 0.131 (0.566) | 0.171 (0.54) | 0.274 (0.522) | 0.216 (0.547)
  Day 90: number analyzed (Participants) | 143 | 117 | 118 | 121 | 128 | 119
  Day 90 | 0.307 (0.609) | 0.184 (0.574) | 0.153 (0.516) | 0.164 (0.579) | 0.275 (0.58) | 0.245 (0.574)
  Follow-up: number analyzed (Participants) | 164 | 131 | 139 | 134 | 145 | 137
  Follow-up | 0.117 (0.621) | 0.226 (0.694) | 0.054 (0.623) | 0.05 (0.572) | 0.175 (0.559) | 0.036 (0.556)

10. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure at Specified Visits
Time Frame: Baseline,Day 7,14,30,60,90,Premature discontinuation (only for participants who have discontinued the study prematurely, to be performed as soon as possible after withdrawal of study drug) and Follow-up (30 days post-last dose, assessed up to Day 120)
Population: Participants in SAF with valid data at specified visits
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 218 | 171 | 160 | 165 | 169 | 163
millimeter of mercury (mmHg)
  Baseline | 120.554 (18.706) | 119.492 (16.348) | 118.498 (14.355) | 119.087 (16.677) | 116.024 (16.895) | 116.941 (16.548)
  Day 7: number analyzed (Participants) | 204 | 158 | 154 | 158 | 163 | 157
  Day 7 | -0.541 (13.894) | -3.178 (13.72) | -2.565 (12.278) | 0.568 (12.733) | 0.162 (15.416) | -0.546 (13.498)
  Day 14: number analyzed (Participants) | 49 | 27 | 40 | 36 | 37 | 32
  Day 14 | -3.442 (14.258) | -4.488 (10.31) | 4.142 (15.001) | 1.241 (13.561) | -3.099 (12.591) | -2.906 (15.406)
  Day 30: number analyzed (Participants) | 177 | 143 | 138 | 147 | 145 | 139
  Day 30 | 0.067 (15.312) | -0.824 (15.747) | -0.367 (14.984) | 0.374 (14.433) | 1.786 (15.039) | 0.899 (14.608)
  Day 60: number analyzed (Participants) | 155 | 128 | 130 | 129 | 139 | 131
  Day 60 | 0.684 (16.315) | 0.337 (14.176) | -1.249 (13.659) | -1.811 (14.462) | 0.981 (15.525) | 0.667 (14.83)
  Day 90: number analyzed (Participants) | 141 | 119 | 121 | 121 | 131 | 122
  Day 90 | -0.967 (16.408) | 0.922 (15.847) | 0.047 (15.643) | -0.664 (15.018) | 1.216 (17.831) | 0.956 (15.743)
  Premature discontinuation: number analyzed (Participants) | 37 | 24 | 24 | 23 | 25 | 24
  Premature discontinuation | -2.991 (16.456) | -0.41 (13.936) | -2.167 (19.963) | 9.391 (22.378) | -2.32 (11.963) | -0.028 (15.42)
  Follow-up: number analyzed (Participants) | 165 | 131 | 141 | 135 | 153 | 143
  Follow-up | 0.188 (16.751) | 2.869 (15.502) | 1.95 (16.148) | -0.928 (17.953) | 2.041 (16.189) | 3.037 (16.782)

11. Other Pre Specified Outcome: Change From Baseline in Diastolic Blood Pressure at Specified Visits
Time Frame: as for outcome 10
Population: Participants in SAF with valid data at specified visits
Measure: Mean (Standard Deviation); unit: millimeter for mercury (mmHg)
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 218 | 171 | 160 | 165 | 169 | 163
millimeter for mercury (mmHg)
  Baseline | 71.633 (11.647) | 71.044 (10.762) | 71.442 (8.508) | 70.61 (9.692) | 70.343 (10.394) | 71.145 (9.809)
  Day 7: number analyzed (Participants) | 204 | 158 | 154 | 158 | 163 | 157
  Day 7 | -1.351 (10.237) | -1.693 (9.911) | -2.143 (9.848) | 0.013 (9.733) | -0.738 (10.534) | -1.166 (8.964)
  Day 14: number analyzed (Participants) | 49 | 27 | 40 | 36 | 37 | 32
  Day 14 | -3.442 (10.089) | -0.537 (9.59) | 1.608 (9.423) | -0.083 (7.421) | -2.387 (10.51) | -0.625 (9.41)
  Day 30: number analyzed (Participants) | 177 | 143 | 138 | 147 | 145 | 139
  Day 30 | -0.503 (10.826) | 0.146 (10.667) | -0.845 (8.91) | -0.068 (9.633) | -0.094 (10.086) | -1.163 (9.622)
  Day 60: number analyzed (Participants) | 155 | 128 | 130 | 129 | 139 | 131
  Day 60 | -0.613 (11.096) | -0.199 (11.297) | -2.144 (9.552) | -0.85 (10.472) | 0.17 (10.312) | -0.575 (10.427)
  Day 90: number analyzed (Participants) | 141 | 119 | 121 | 121 | 131 | 122
  Day 90 | -0.716 (11.035) | -0.106 (11.148) | -1.738 (9.015) | -1.121 (9.96) | -0.545 (11.212) | -0.877 (11.327)
  Premature discontinuation: number analyzed (Participants) | 36 | 24 | 24 | 23 | 25 | 24
  Premature discontinuation | -3.185 (11.853) | 0.868 (9.239) | -2.194 (15.522) | 4.101 (12.151) | -2.96 (9.199) | -0.083 (10.113)
  Follow-up: number analyzed (Participants) | 165 | 131 | 141 | 135 | 153 | 143
  Follow-up | -1.218 (11.477) | 0.696 (13.172) | -0.444 (10.197) | -1.16 (11.114) | -0.298 (11.521) | -0.172 (10.211)

12. Other Pre Specified Outcome: Change From Baseline in Heart Rate at Specified Visits
Time Frame: as for outcome 10
Population: Participants in SAF with valid data at specified visits
Measure: Mean (Standard Deviation); unit: Beats per minute (Beats/min)
Arm/Group | Eplerenone (INSPRA®) | Finerenone (BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
Number analyzed (Participants) | 217 | 171 | 160 | 165 | 169 | 162
Beats per minute (Beats/min)
  Baseline | 74.957 (13.813) | 73.369 (13.396) | 72.681 (12.623) | 74.184 (12.369) | 73.852 (11.999) | 74.329 (13.187)
  Day 7: number analyzed (Participants) | 203 | 158 | 153 | 158 | 163 | 157
  Day 7 | -0.8 (10.751) | 1.073 (13.5) | -0.63 (11.696) | -0.719 (10.77) | -0.548 (11.144) | -1.176 (13.398)
  Day 14: number analyzed (Participants) | 49 | 27 | 40 | 36 | 37 | 32
  Day 14 | -3.109 (15.101) | 0.599 (16.387) | 1.842 (14.988) | -1.324 (13.666) | 0.423 (11.247) | -3.969 (13.715)
  Day 30: number analyzed (Participants) | 176 | 143 | 138 | 147 | 145 | 139
  Day 30 | 0.294 (13.61) | 1.064 (14.128) | 0.435 (13.63) | -0.349 (12.636) | -0.802 (11.311) | -1.633 (12.719)
  Day 60: number analyzed (Participants) | 155 | 128 | 130 | 129 | 139 | 131
  Day 60 | 0.297 (13.033) | -0.975 (14.953) | -1.741 (10.86) | -2.318 (14.225) | 0.192 (13.377) | -1.608 (13.828)
  Day 90: number analyzed (Participants) | 141 | 119 | 121 | 121 | 131 | 122
  Day 90 | -0.189 (12.289) | -1.647 (13.001) | -2.89 (12.034) | -2.212 (12.041) | -0.71 (13.777) | -1.145 (14.284)
  Premature discontinuation: number analyzed (Participants) | 36 | 24 | 24 | 23 | 25 | 23
  Premature discontinuation | -2.278 (15.909) | -1.424 (15.587) | -0.222 (7.591) | 1.101 (10.22) | 4.733 (13.646) | -2.072 (19.731)
  Follow-up: number analyzed (Participants) | 165 | 131 | 141 | 135 | 153 | 143
  Follow-up | -1.281 (13.789) | -2.057 (13.982) | -0.626 (14.196) | -1.326 (15.488) | 0.834 (14.159) | -1.317 (14.636)

ADVERSE EVENTS:
Time Frame: Adverse events: from the start of study treatment until 3 days post-last dose, up to approximately 93 days. All Cause Mortality: assessed until 30 days post-last dose, up to approximately 120 days.
Groups:
- Finerenone(BAY94-8862) 2.5-5 mg OD: Finerenone 2.5 mg immediate-release (IR) tablets OD and placebo-matched to Eplerenone capsule OD, with possible up-titration to 5 mg OD at Day 30 (Day 30±2) and sham up-titration at Day 60 (Day 60±2). Treatment duration was for 90 days.
Arm/Group | Eplerenone (INSPRA®) | Finerenone(BAY94-8862) 2.5-5 mg OD | Finerenone (BAY94-8862) 5-10 mg OD | Finerenone (BAY94-8862) 7.5-15 mg OD | Finerenone (BAY94-8862) 10-20 mg OD | Finerenone (BAY94-8862) 15-20 mg OD
All-Cause Mortality (participants affected / at risk) | 19/221 | 17/172 | 9/163 | 12/167 | 2/169 | 9/163
Serious Adverse Events (participants affected / at risk) | 77/221 | 72/172 | 47/163 | 52/167 | 46/169 | 57/163
Other Adverse Events (participants affected / at risk) | 85/221 | 63/172 | 59/163 | 50/167 | 50/169 | 65/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (INSPRA®) (N=221) | Finerenone(BAY94-8862) 2.5-5 mg OD (N=172) | Finerenone (BAY94-8862) 5-10 mg OD (N=163) | Finerenone (BAY94-8862) 7.5-15 mg OD (N=167) | Finerenone (BAY94-8862) 10-20 mg OD (N=169) | Finerenone (BAY94-8862) 15-20 mg OD (N=163)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 21 (27) | 16 (26) | 15 (17) | 21 (33) | 11 (12) | 13 (14)
Cardiac failure acute (Cardiac disorders) | 6 (6) | 6 (6) | 3 (3) | 1 (1) | 3 (4) | 5 (5)
Cardiac failure chronic (Cardiac disorders) | 13 (16) | 9 (11) | 7 (7) | 8 (9) | 6 (6) | 12 (16)
Cardiac failure congestive (Cardiac disorders) | 4 (5) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 3 (7)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 4 (8) | 0 (0) | 3 (5) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema due to cardiac disease (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Implant site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implant site ulcer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent-graft endoleak (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Computerised tomogram abdomen abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 6 (6) | 4 (4) | 7 (7) | 5 (5) | 6 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 5 (5) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac pacemaker removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardioversion (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toe amputation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Implantable defibrillator insertion (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular assist device insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac resynchronisation therapy (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemodynamic instability (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eplerenone (INSPRA®) (N=221) | Finerenone(BAY94-8862) 2.5-5 mg OD (N=172) | Finerenone (BAY94-8862) 5-10 mg OD (N=163) | Finerenone (BAY94-8862) 7.5-15 mg OD (N=167) | Finerenone (BAY94-8862) 10-20 mg OD (N=169) | Finerenone (BAY94-8862) 15-20 mg OD (N=163)
Cardiac failure (Cardiac disorders) | 13 (14) | 14 (20) | 10 (11) | 5 (6) | 7 (7) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 6 (6) | 6 (6) | 10 (11) | 6 (6) | 7 (9)
Nausea (Gastrointestinal disorders) | 7 (7) | 9 (12) | 2 (2) | 5 (7) | 2 (2) | 6 (6)
Blood creatinine increased (Investigations) | 12 (14) | 5 (5) | 7 (7) | 3 (3) | 4 (4) | 8 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 8 (9) | 5 (5) | 7 (10) | 7 (7) | 6 (6) | 9 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 34 (44) | 20 (26) | 21 (28) | 15 (30) | 14 (18) | 17 (20)
Dizziness (Nervous system disorders) | 12 (13) | 8 (8) | 6 (7) | 6 (6) | 7 (7) | 6 (7)
Renal impairment (Renal and urinary disorders) | 8 (10) | 6 (8) | 7 (9) | 6 (10) | 8 (11) | 9 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 12 (13) | 7 (7) | 6 (7) | 3 (4) | 10 (11)
Hypotension (Vascular disorders) | 11 (13) | 7 (7) | 11 (12) | 11 (14) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other